CLINICAL TRIAL: NCT00000362
Title: Randomized Study of Two Interventions for Liquid Aspiration: Short-Term and Long-Term Effects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIDCD-1159; Protocol 201; U01DC003206 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2006-04-24 (Estimated); Status verified 2006-04

CONDITIONS: Pneumonia, Aspiration
Keywords: Deglutition Disorders; Dementia; Parkinson Disease; Pneumonia, Aspiration
MeSH Terms: conditions — Pneumonia, Aspiration; Deglutition Disorders; Dementia; Parkinson Disease

INTERVENTIONS:
Behavioral: Chin-down position
Behavioral: Thickened liquid administration

SUMMARY:
The purpose of this study is to determine whether chin-down posture or use of a thickened liquid diet is more effective in the prevention of aspiration and aspiration pneumonia in patients with Parkinson's disease and/or dementia. Liquid aspiration is the most common type of aspiration in older populations, especially those suffering from debilitation, dementia, and depression. Pneumonia may develop as a consequence of aspiration and is the fifth leading cause of death in the US among persons age 65 years and over. Current treatment involves either use of chin-down position with swallowing or use of thickened liquids in the diet, without any clear evidence supporting the use of one treatment over the other. This is a Phase III inpatient and/or outpatient study in which all participants will be randomly assigned to either the chin-down position or the thickened liquid treatment group based on swallowing function during a modified barium swallow. This study is scheduled to recruit patients for a three-year period; participation by each individual patient spans no more than three months after entry.

ELIGIBILITY:
Inclusion Criteria:

* Have dementia or Parkinson's disease and are found to aspirate on thin liquid during a set of qualifying swallows.

Exclusion Criteria:

* Have smoked more than a pack of cigarettes per day in the last year.
* Drink more than 3 alcoholic beverages per day on a regular basis.
* Have had any head and neck cancer treatment.
* Have any head and neck anatomic deformities.
* Have a history of 20 years or longer of insulin-dependent diabetes.
* Have other exclusionary neurologic diagnoses.
* Have had pneumonia within 6 weeks of screening.
* Currently have a nasogastric tube.
* Currently have a tracheotomy.
* Are a resident in non-participating nursing home or assisted living environment.
* Live alone.
* Have no regular care provider present at meals.
* Have no Speech-Language Pathologist to provide a 3-month follow-up.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Joanne Robbins, Study Chair; Dr. Jeri Logemann, Principal Investigator
Locations (1):
- University of Wisconsin at Madison & multiple other U.S. locations, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Robbins J, Gensler G, Hind J, Logemann JA, Lindblad AS, Brandt D, Baum H, Lilienfeld D, Kosek S, Lundy D, Dikeman K, Kazandjian M, Gramigna GD, McGarvey-Toler S, Miller Gardner PJ. Comparison of 2 interventions for liquid aspiration on pneumonia incidence: a randomized trial. Ann Intern Med. 2008 Apr 1;148(7):509-18. doi: 10.7326/0003-4819-148-7-200804010-00007. PMID 18378947